CLINICAL TRIAL: NCT07319299
Title: A Prospective, Interventional, Longitudinal APAC Study Evaluating Clinical Utility of GAAD Score for Detection of Hepatocellular Carcinoma in a High-risk APAC Patient Population
Brief Title: STOP HCC-GAAD-APAC-Thailand
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Si 089/2024
Record Dates: First submitted 2025-11-15; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Hepatecellular Carcinoma; Cirrhosis; HBV Infection
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Intervention Model Description: GAAD score
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GAAD Score (Other): All enrolled participants will undergo standard hepatocellular carcinoma (HCC) surveillance consisting of blood sampling and abdominal ultrasound performed every 6 months for a total follow-up period of 24 months. Blood samples will be analyzed for serum alpha-fetoprotein (AFP) and protein induced by vitamin K absence or antagonist-II (PIVKA-II) to calculate the GAAD score, a multivariable index incorporating gender, age, AFP, and PIVKA-II.
  A GAAD score ≥ 2.57 will trigger a recall procedure, defined as diagnostic evaluation with multiphasic contrast-enhanced computed tomography (CT) or magnetic resonance imaging (MRI) of the liver. This recall procedure is conducted in addition to standard surveillance recall criteria, which include detection of a suspicious hepatic lesion measuring ≥ 1 cm on ultrasound or elevated or rising serum AFP levels (≥ 20 ng/mL).
  Interventions: Diagnostic Test: GAAD score

INTERVENTIONS:
Diagnostic Test: GAAD score — All enrolled participants will undergo standard hepatocellular carcinoma (HCC) surveillance, consisting of blood sampling and abdominal ultrasound performed every 6 months for a total follow-up period of 24 months. Blood samples will be analyzed for serum alpha-fetoprotein (AFP) and protein induced by vitamin K absence or antagonist-II (PIVKA-II) to calculate the GAAD score, a multivariable index incorporating gender, age, AFP, and PIVKA-II.
  A GAAD score of ≥ 2.57 will trigger a recall procedure, defined as further diagnostic evaluation using multiphasic contrast-enhanced computed tomography (CT) or magnetic resonance imaging (MRI) of the liver. This recall procedure is performed in addition to standard surveillance recall criteria, which include detection of a suspicious hepatic lesion measuring ≥ 1 cm on ultrasound or elevated or rising serum AFP levels (≥ 20 ng/mL).

SUMMARY:
Hepatocellular carcinoma (HCC) surveillance is frequently underutilized, and currently available biomarkers, such as alpha-fetoprotein (AFP), demonstrate suboptimal diagnostic performance. This prospective study aims to evaluate a simplified multivariate index, the GAAD score-comprising gender, age, alpha-fetoprotein (AFP), and protein induced by vitamin K absence or antagonist-II (PIVKA-II)-for its ability to improve the detection of hepatocellular carcinoma in patients with chronic liver disease.

The study hypothesizes that incorporation of the GAAD score into standard HCC surveillance strategies will improve diagnostic performance compared with existing surveillance modalities alone and may provide evidence to support its inclusion in future clinical practice guidelines.

DETAILED DESCRIPTION:
Surveillance and early detection of hepatocellular carcinoma (HCC) increase the likelihood of potentially curative treatment. However, HCC surveillance remains substantially underutilized, even in countries with adequate healthcare resources. Early-stage HCC can be treated with curative intent using local ablation, surgical resection, or liver transplantation.

The role of serum alpha-fetoprotein (AFP) in HCC surveillance varies across international guidelines. AFP is recommended for surveillance by the Asian Pacific Association for the Study of the Liver (APASL), considered optional by the American Association for the Study of Liver Diseases (AASLD), and not recommended by the European Association for the Study of the Liver (EASL). Similar considerations have informed recommendations for combined use of AFP with ultrasound (US) in HCC surveillance by the World Health Organization (WHO) Guidelines for the Prevention, Care and Treatment of Viral Hepatitis (references 1-4).

AFP has demonstrated suboptimal performance as a serologic surveillance marker for HCC. Serum AFP levels may fluctuate in patients with cirrhosis due to hepatitis B virus (HBV) or hepatitis C virus (HCV) activity, exacerbations of underlying liver disease, or the development of HCC, thereby limiting its diagnostic accuracy.

Recently, the GALAD score-a multivariable model incorporating gender, age, AFP-L3, AFP, and protein induced by vitamin K absence or antagonist-II (PIVKA-II)-has been proposed as an alternative approach to improve HCC detection and has demonstrated strong diagnostic performance in patients with cirrhotic HCC. A simplified version of this model, the GAAD score (Roche Diagnostics International Ltd., Rotkreuz, Switzerland), which includes gender, age, AFP, and PIVKA-II, has been shown to achieve comparable diagnostic performance in preliminary analyses (Piratvisuth et al., 2023, submitted).

However, the existing evidence supporting the use of the GALAD and GAAD scores is primarily derived from retrospective and/or case-control studies. Prospective validation in real-world surveillance settings remains limited. This study is therefore designed to prospectively evaluate the diagnostic performance of the GAAD score, alone and in combination with standard surveillance modalities, in patients with chronic liver disease undergoing routine HCC surveillance.

ELIGIBILITY:
Inclusion Criteria:

* Adults with chronic liver disease who have an indication for hepatocellular carcinoma (HCC) surveillance, including one or more of the following:
* Liver cirrhosis of any etiology (e.g., chronic hepatitis B virus [HBV], chronic hepatitis C virus [HCV], metabolic dysfunction-associated steatohepatitis [MASH], or alcohol-related liver disease [ALD])
* Non-cirrhotic chronic liver disease (e.g., HCV, MASH, or ALD) with evidence of stage F3 fibrosis
* Chronic HBV infection with a clinical diagnosis of non-cirrhotic liver disease

Exclusion Criteria:

* Diagnosis of any active malignancy other than non-melanoma skin cancer
* History of previously diagnosed malignancy, including prior hepatocellular carcinoma
* Life expectancy of less than 2 years
* Use of vitamin K antagonists within 1 week prior to enrollment
* Pregnant or breastfeeding women
* Estimated glomerular filtration rate (GFR) < 60 mL/min/1.73 m²
* Significant hepatic decompensation or Child-Pugh class C liver disease
* Unwillingness or inability to undergo computed tomography (CT) or magnetic resonance imaging (MRI)
* Unwillingness or inability to provide informed consent or to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2100 (Estimated)
Dates: Start 2025-02-02 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
True Positive Rate (Sensitivity) of Ultrasound, AFP, and GAAD Score as Standalone Surveillance Modalities | Over 24 months of patient follow-up
  To evaluate the true positive rate (sensitivity) of Ultrasound, serum alpha-fetoprotein (AFP), and the GAAD score when used individually for hepatocellular carcinoma (HCC) surveillance. Sensitivity will be calculated for each modality separately by comparing surveillance results with the reference standard diagnosis of HCC. Unit of Measure: Proportion (percentage)
False Positive Rate of Ultrasound, AFP, and GAAD Score as Standalone Surveillance Modalities | Over 24 months of patient follow-up
  To evaluate the false positive rate of Ultrasound, serum AFP, and the GAAD score when used individually for HCC surveillance. The false positive rate will be calculated for each modality separately based on surveillance results compared with the reference standard diagnosis. Unit of Measure: Proportion (percentage)
True Positive Rate (Sensitivity) of Combined Ultrasound + GAAD Score for HCC Surveillance | Over 24 months of patient follow-up
  To evaluate the true positive rate (sensitivity) of the combined Ultrasound and GAAD score strategy for HCC surveillance. A positive surveillance result will be defined according to the prespecified combination criteria (e.g., either test positive or both tests positive, as defined in the protocol). Unit of Measure: Proportion (percentage)
False Positive Rate of Combined Ultrasound + GAAD Score for HCC Surveillance | Over 24 months of patient follow-up
  To evaluate the false positive rate of the combined Ultrasound and GAAD score strategy for HCC surveillance, using the reference standard diagnosis of HCC. Unit of Measure: Proportion (percentage)
True Positive Rate (Sensitivity) of Combined Ultrasound + AFP for HCC Surveillance | Over 24 months of patient follow-up
  To evaluate the true positive rate (sensitivity) of the combined Ultrasound and serum AFP strategy for HCC surveillance, based on predefined combination criteria. Unit of Measure: Proportion (percentage)
False Positive Rate of Combined Ultrasound + AFP for HCC Surveillance | Over 24 months of patient follow-up
  To evaluate the false positive rate of the combined Ultrasound and serum AFP strategy for HCC surveillance, compared with the reference standard diagnosis of HCC. Unit of Measure: Proportion (percentage)

SECONDARY OUTCOMES:
Area Under the Receiver Operating Characteristic Curve (AUC) of GAAD Compared With Ultrasound, AFP, and PIVKA-II | Over 24 months of patient follow-up
  o compare the overall discriminative ability of the GAAD algorithm with Ultrasound, serum AFP, and serum PIVKA-II for the detection of hepatocellular carcinoma (HCC). Performance will be assessed using the area under the receiver operating characteristic curve (AUC), stratified by HCC stage and underlying liver disease etiology. Unit of Measure: AUC (unitless)
Sensitivity and Specificity of GAAD Compared With Ultrasound, AFP, and PIVKA-II | Over 24 months of patient follow-up
  To compare the sensitivity and specificity of the GAAD algorithm with Ultrasound, serum AFP, and serum PIVKA-II for HCC surveillance. Sensitivity and specificity will be calculated separately for each modality and stratified by HCC stage and etiology. Unit of Measure: Proportion (percentage)
Positive Predictive Value (PPV) and Negative Predictive Value (NPV) of GAAD Compared With Ultrasound, AFP, and PIVKA-II | Over 24 months of patient follow-up
  To compare the positive predictive value (PPV) and negative predictive value (NPV) of the GAAD algorithm with Ultrasound, serum AFP, and serum PIVKA-II for HCC surveillance, stratified by HCC stage and etiology. Unit of Measure: Proportion (percentage)
Area Under the Receiver Operating Characteristic Curve (AUC) of Combined Ultrasound + AFP | Over 24 months of patient follow-up
  To evaluate the discriminative performance of the combined Ultrasound and serum AFP strategy for HCC surveillance using the area under the receiver operating characteristic curve (AUC), stratified by HCC stage and etiology. Unit of Measure: AUC (unitless)
Sensitivity and Specificity of Combined Ultrasound + AFP | Over 24 months of patient follow-up
  To evaluate the sensitivity and specificity of the combined Ultrasound and serum AFP strategy for HCC surveillance, stratified by HCC stage and etiology. Unit of Measure: Proportion (percentage)
Positive Predictive Value (PPV) and Negative Predictive Value (NPV) of Combined Ultrasound + AFP | Over 24 months of patient follow-up
  To evaluate the positive predictive value (PPV) and negative predictive value (NPV) of the combined Ultrasound and serum AFP strategy for HCC surveillance, stratified by HCC stage and etiology. Unit of Measure: Proportion (percentage)
Longitudinal Changes in AFP Levels Prior to HCC Diagnosis | Over 24 months of patient follow-up
  To assess longitudinal changes in serum Elecsys AFP concentrations preceding an HCC diagnosis among confirmed HCC cases. Unit of Measure: Nanograms per milliliter (ng/mL)
Longitudinal Changes in PIVKA-II Levels Prior to HCC Diagnosis | Over 24 months of patient follow-up
  To assess longitudinal changes in serum Elecsys PIVKA-II concentrations preceding an HCC diagnosis among confirmed HCC cases. Unit of Measure: milli-arbitrary units per milliliter (mAU/mL)
Longitudinal Changes in GAAD Score Prior to HCC Diagnosis | Over 24 months of patient follow-up
  To assess longitudinal changes in the GAAD score preceding an HCC diagnosis among confirmed HCC cases. Unit of Measure: Unitless score
Number of Additional Early-Stage HCCs Detected Using GAAD | Over 24 months of patient follow-up
  To quantify the number of additional early-stage hepatocellular carcinoma cases identified using the GAAD score compared with standard surveillance modalities. Unit of Measure: Number of participants
Number of Additional CT or MRI Imaging Procedures Triggered by Surveillance Tests | Over 24 months of patient follow-up
  To count the number of additional CT or MRI imaging procedures triggered by positive results from GAAD, AFP, or Ultrasound surveillance tests. Unit of Measure: Number of imaging procedures
Relative False Positive Rate of Additional CT or MRI Imaging Procedures | Over 24 months of patient follow-up
  To calculate the relative false positive rate of additional CT or MRI imaging procedures triggered by positive GAAD, AFP, or Ultrasound surveillance results. Unit of Measure: Proportion (percentage)

CONTACTS AND LOCATIONS:
Overall Officials: Tawesak Tanwandee, MD, Principal Investigator — Siriraj Hospital; Tawesak Tanwandee, MD, Study Director — Siriraj Hospital; Tawesak Tanwandee, MD, Study Chair — Siriraj Hospital; Tawesak Tanwandee, Principal Investigator — Siriraj Hospital
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
The datasets generated and/or analysed during the current study are not publicly available due to the policy of the institutes.

REFERENCES:
- [Result] Tzartzeva K, Obi J, Rich NE, Parikh ND, Marrero JA, Yopp A, Waljee AK, Singal AG. Surveillance Imaging and Alpha Fetoprotein for Early Detection of Hepatocellular Carcinoma in Patients With Cirrhosis: A Meta-analysis. Gastroenterology. 2018 May;154(6):1706-1718.e1. doi: 10.1053/j.gastro.2018.01.064. Epub 2018 Feb 6. PMID 29425931
- [Result] Best J, Bechmann LP, Sowa JP, Sydor S, Dechene A, Pflanz K, Bedreli S, Schotten C, Geier A, Berg T, Fischer J, Vogel A, Bantel H, Weinmann A, Schattenberg JM, Huber Y, Wege H, von Felden J, Schulze K, Bettinger D, Thimme R, Sinner F, Schutte K, Weiss KH, Toyoda H, Yasuda S, Kumada T, Berhane S, Wichert M, Heider D, Gerken G, Johnson P, Canbay A. GALAD Score Detects Early Hepatocellular Carcinoma in an International Cohort of Patients With Nonalcoholic Steatohepatitis. Clin Gastroenterol Hepatol. 2020 Mar;18(3):728-735.e4. doi: 10.1016/j.cgh.2019.11.012. Epub 2019 Nov 8. PMID 31712073
- [Result] Omata M, Cheng AL, Kokudo N, Kudo M, Lee JM, Jia J, Tateishi R, Han KH, Chawla YK, Shiina S, Jafri W, Payawal DA, Ohki T, Ogasawara S, Chen PJ, Lesmana CRA, Lesmana LA, Gani RA, Obi S, Dokmeci AK, Sarin SK. Asia-Pacific clinical practice guidelines on the management of hepatocellular carcinoma: a 2017 update. Hepatol Int. 2017 Jul;11(4):317-370. doi: 10.1007/s12072-017-9799-9. Epub 2017 Jun 15. PMID 28620797
- [Result] European Association for the Study of the Liver. EASL Clinical Practice Guidelines: Management of hepatocellular carcinoma. J Hepatol. 2018 Jul;69(1):182-236. doi: 10.1016/j.jhep.2018.03.019. Epub 2018 Apr 5. No abstract available. Erratum In: J Hepatol. 2019 Apr;70(4):817. doi: 10.1016/j.jhep.2019.01.020. PMID 29628281
- [Result] Singal AG, Llovet JM, Yarchoan M, Mehta N, Heimbach JK, Dawson LA, Jou JH, Kulik LM, Agopian VG, Marrero JA, Mendiratta-Lala M, Brown DB, Rilling WS, Goyal L, Wei AC, Taddei TH. AASLD Practice Guidance on prevention, diagnosis, and treatment of hepatocellular carcinoma. Hepatology. 2023 Dec 1;78(6):1922-1965. doi: 10.1097/HEP.0000000000000466. Epub 2023 May 22. No abstract available. PMID 37199193

DOCUMENTS (1):
  • Study Protocol (2025-10-17): https://cdn.clinicaltrials.gov/large-docs/99/NCT07319299/Prot_000.pdf